CLINICAL TRIAL: NCT01208805
Title: Spinal Cord Evoked Potentials in Candidates for Dorsal Column Stimulation
Brief Title: Spinal Cord Evoked Potentials as a Tool to Investigate Sensorimotor Processing
Acronym: SCEPTISM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Prof Bart Nuttin, UZ Leuven
Other Study IDs: S52573
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Studying Spinal Cord Evoked Potentials in Patients With Intractable Pain.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Candidates for dorsal column stimulation
  Interventions: Behavioral: Recording spinal cord evoked potentials

INTERVENTIONS:
Behavioral: Recording spinal cord evoked potentials — Recording spinal cord evoked potentials from patients suffering from intractable pain in whom epidural electrodes have already been implanted

SUMMARY:
The study first aim is to investigate the relationship between different patterns of electrode stimulation and peripheral sensory stimulation and spinal cord-evoked potentials to optimize spinal cord stimulation parameters . The second aim of the study is to investigate the role of the spinal cord in some aspects of cognitive-sensory-motor processing, specifically the presence of top-down attentional effects on the sensory analysis of an external stimulus at the spinal cord level.

The study will be performed on patients that will be implanted with a spinal epidural electrode because of chronic intractable pain. From these electrodes, spinal cord evoked potentials (SCEPs) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 70
* Candidates for spinal cord stimulation
* Epidural electrode at the the level of the cervical or thoracic spine.

Exclusion Criteria:

* Generalized sensory deficit interfering with the recording of spinal cord evoked potentials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with epidural elektrodes for intractable pain (spinal cord stimulation)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-12 (Estimated); Study Completion 2012-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Brabant, Belgium